CLINICAL TRIAL: NCT03882606
Title: Near Visual Acuity and Quality of Life Improvement After Implantation of the add-on Scharioth Macula Lens (SML, Medicontur) in Patients With Dry Age-related Macular Degeneration and Myopic Maculopathy
Brief Title: Implantation of SML in Patients With Dry Age-related Macular Degeneration and Myopic Maculopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Consorci Sanitari de Terrassa (Other)
Collaborators: Medicontur Medical Engineering Ltd (Industry)
Responsible Party: Principal Investigator, Laura Gutiérrez-Benítez, MD, Consorci Sanitari de Terrassa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GUTSML201902
Record Dates: First submitted 2019-02-22; First posted 2019-03-20 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2023-09

CONDITIONS: Age-Related Macular Degeneration; Lens, Intraocular; Myopic Maculopathy
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- SML implantation (Other): prospective study of a cohort of patients with age-related macular degeneration or myopic maculopathy treated with SML implantation
  Interventions: Device: Scharioth Macula Lens (SML, Medicontur)

INTERVENTIONS:
Device: Scharioth Macula Lens (SML, Medicontur) — magnifying intraocular lens for pseudophakic patients implanted in the ciliary sulcus in one eye of each patient

SUMMARY:
Age-related macular degeneration (AMD) is the leading cause of irreversible vision loss in developed countries among people over 50 years of age. Myopic maculopathy is also an important cause of irreversible vision loss. Reduced near visual acuity is still a major problem with all forms of AMD and myopic maculopathy. Various intraocular lenses for near vision (IOLs) or telescopic systems have been described but are not widely accepted and almost all solutions require phakic status of the eye and are implanted during cataract surgery. Therefore, these devices are not appropriated for pseudophakic AMD and myopic maculopathy patients. Scharioth Macula Lens (SML, Medicontur) is a magnifying intraocular lens for pseudophakic patients implanted in the ciliary sulcus in one eye of each patient. The implant has a bifocal optic, with a central 1.5mm diameter optical zone equivalent to +10D add and a peripheral zone optically neutral. The implantation of the add-on SML can improve the near visual acuity of pseudophakic patients with AMD and myopic maculopathy without impairing their distance visual acuity.

The principal objective is to compare the near visual acuity, the far visual acuity and the self-reported vision health status before and after the SML implantation.

DETAILED DESCRIPTION:
We present a prospective study of a cohort of patients with age-related macular degeneration and myopic maculopathy treated with SML implantation. The study was approved by the ethics committee at the Consorci Sanitari de Terassa (Barcelona, Spain).

Patients will be examined for best corrected visual acuity prior to the surgery at 6 meter and for reading at 40cm (with a +2.5D) and 15 cm (with +6D). Improvement of the reading ability at 15 cm compared to 40 cm will predict the potential for vision improvement with the add on lens.

The preoperative and postoperative assessment will include a full ophthalmological exam, visual acuity for distance and near, optical coherence tomography of the anterior chamber and of the macula, axial length and keratometry examination using biometry and VFQ25 questionnaire.

Postoperative assessment will be performed at day 1, 1 week, 1, 3 and 6 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Eye with better distance visual acuity or non-dominant eye in case of equal visual acuity in both eyes
* Best corrected visual acuity 0.1-0.4 (Snellen)
* Pseudophakia
* Preoperative testing of corrected near visual acuity (CNVA) at 15cm (+6 D) better than CNVA at 40 cm (+2.5D)
* understand the principle of this implant (reduced reading distance, maximum magnification)
* signing the informed consent

Exclusion Criteria:

* complicated cataract surgery
* excessive zonular weakness
* chronic uveitis
* active rubeosis iridis
* central corneal opacities
* inability to understand the principle of this implant (reduced reading distance, maximum magnification)
* Narrow anterior chamber (<2.8mm)
* Narrow angle
* glaucoma
* Phakic
* Current treatment with intravitreal injections
* active maculopathy
* atrophy
* photopic pupil size less than 2.5 mm
* severe eye pathology
* previous retinal surgery

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2019-05-22 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
change in near visual acuity | will be performed at day 1, 1 week, 1, 3 and 6 months after surgery
  to compare the near visual acuity before and after the SML implantation
change in VFQ25 score | will be performed at day 1, 1 week, 1, 3 and 6 months after surgery
  to compare the VFQ25 score before and after the SML implantation
change in far visual acuity | will be performed at day 1, 1 week, 1, 3 and 6 months after surgery
  to compare the far visual acuity before and after the SML implantation

CONTACTS AND LOCATIONS:
Locations (1):
- Consorci Sanitari de Terrassa, Terrassa, Barcelona (spain), Spain

IPD SHARING:
Plan to Share IPD: No